CLINICAL TRIAL: NCT00883090
Title: A 12 Week, Multicenter, Pharmacokinetic and Safety Study of Human Plasma-Derived Factor XIII Concentrate in Subjects With Congenital Factor XIII Deficiency
Brief Title: A Study of the Use of Factor XIII Concentrate in Patients With Inherited FXIII Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BI71023_2002; 2009-010387-41 (EudraCT Number); 1479 (Other: CSL Behring)
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2011-12

CONDITIONS: Factor XIII Deficiency
Keywords: Factor XIII
MeSH Terms: conditions — Factor XIII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FXIII (Experimental): All subjects treated with Factor XIII Concentrate (Human) (FXIII)
  Interventions: Biological: FXIII Concentrate (Human)

INTERVENTIONS:
Biological: FXIII Concentrate (Human) — Subjects will receive approximately 40 U/kg of FXIII every 28 days for 3 doses administered as a bolus intravenous (IV) injection at approximately 250 U/minute.
  Other Names: Fibrogammin®-P

SUMMARY:
Congenital deficiency of Factor XIII is an extremely rare hereditary disorder associated with potentially life-threatening bleeding. This study will evaluate the safety and recommended (best) amount or level of Factor XIII in a patient's blood. Factor XIII Concentrate (Human) is given to people whose blood is lacking Factor XIII. Factor XIII Concentrate (Human) works by assisting your blood in the usual clotting process, thereby preventing bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent for study participation obtained before undergoing any study-specific procedures
* Documented congenital FXIII deficiency that requires prophylactic treatment with a FXIII containing product.
* Males and females of any age with congenital FXIII deficiency.
* Received full hepatitis B vaccination and/or is hepatitis B surface antibody positive

Exclusion Criteria:

* Diagnosis of acquired FXIII deficiency
* Administration of a FXIII-containing product, including blood transfusions or other blood products within 4 weeks prior to the planned Day 0
* Any known congenital or acquired coagulation disorder other than congenital FXIII deficiency
* Known or suspected to have antibodies towards FXIII
* Use of any other investigational medicinal product within 4 weeks prior to the Baseline Visit (Day 0)
* Positive result at screening for human immunodeficiency virus (HIV)
* Serum aspartate transaminase (AST) or serum alanine transaminase (ALT) concentration >2.5 times the upper limit of normal
* Fibrinogen < lower limit of normal
* Active bleeding
* Pregnant or breast-feeding
* Intention to become pregnant during the course of the study
* Female subjects of childbearing potential not using, or not willing to use, a medically reliable method of contraception for the entire duration of the study
* Surgical procedure anticipated during the study period
* Suspected inability (e.g., language problems) or unwillingness to comply with study procedures or history of noncompliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (6):
- United States (5):
  - Study Site, Dothan, Alabama
  - Study Site, Orange, California
  - Study Site, San Francisco, California
  - Study Site, Stockton, California
  - Study Site, Boston, Massachusetts
- Study Site, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Derived] Nugent DJ, Ashley C, Garcia-Talavera J, Lo LC, Mehdi AS, Mangione A. Pharmacokinetics and safety of plasma-derived factor XIII concentrate (human) in patients with congenital factor XIII deficiency. Haemophilia. 2015 Jan;21(1):95-101. doi: 10.1111/hae.12505. Epub 2014 Dec 2. PMID 25458735

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was not administered FXIII because of the Sponsor's decision. This subject was not included in the analyses.
Period: Overall Study
Arm/Group | FXIII
Started | 15 (Of the 15 participants started, 14 were administered FXIII)
Completed | 13
Not Completed | 2
Not completed — Sponsor's decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- FXIII: All subjects treated with Factor FXIII Concentrate (Human) (FXIII)
Arm/Group | FXIII
Number analyzed (Participants) | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 24.0 (12.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Peak FXIII Concentration at Steady State
Time Frame: 12 weeks
Population: The analysis population was the pharmacokinetic (PK) population. The PK population comprised all subjects in the safety population who completed the study (defined as having sufficient bioanalytical assessments to calculate reliable estimates of the PK parameters specified).
Measure: Mean (Standard Deviation); unit: Units/mL
Arm/Group | FXIII
Number analyzed (Participants) | 13
Units/mL | 0.9 (0.20)

2. Primary Outcome: Trough FXIII Concentration at Steady State
Time Frame: 12 weeks
Population: The analysis population was the PK population. The PK population comprised all subjects in the safety population who completed the study (defined as having sufficient bioanalytical assessments to calculate reliable estimates of the PK parameters specified).
Measure: Mean (Standard Deviation); unit: Units/mL
Arm/Group | FXIII
Number analyzed (Participants) | 13
Units/mL | 0.05 (0.05)

3. Primary Outcome: Time to Peak Concentration
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | FXIII
Number analyzed (Participants) | 13
hr | 1.7 (1.44)

4. Primary Outcome: Incremental Recovery
Description: Incremental recovery (U/mL/U/kg) is defined as the maximum (peak) FXIII activity (U/mL) obtained after infusion, per dose of FXIII (U/kg) administered.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/mL/Units/kg
Arm/Group | FXIII
Number analyzed (Participants) | 13
Units/mL/Units/kg | 0.02 (0.01)

5. Primary Outcome: Terminal Half-life
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FXIII
Number analyzed (Participants) | 13
days | 6.6 (2.29)

6. Primary Outcome: Area Under the Curve at Steady State
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units*hr/mL
Arm/Group | FXIII
Number analyzed (Participants) | 13
Units*hr/mL | 184.0 (65.78)

7. Primary Outcome: Clearance
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | FXIII
Number analyzed (Participants) | 13
mL/hr/kg | 0.25 (0.09)

8. Primary Outcome: Volume of Distribution at Steady State
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | FXIII
Number analyzed (Participants) | 13
mL/kg | 51.1 (12.61)

9. Primary Outcome: Mean Residence Time
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FXIII
Number analyzed (Participants) | 13
days | 10.0 (3.45)

10. Secondary Outcome: Adverse Events
Description: Number of participants with an adverse event
Time Frame: 16 weeks
Population: The analysis population was the safety population. The safety population comprised all subjects who received a dose of Factor XIII.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 14
participants | 8

11. Secondary Outcome: Laboratory Safety Parameters
Description: Number of participants with clinically significant laboratory safety parameter values. The laboratory safety parameters measured included serum chemistries, hematology and urinalysis.
Time Frame: 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 14
participants | 0

12. Secondary Outcome: Vital Signs
Description: Number of participants with clinically significant vital signs. The vital signs measured included blood pressure, pulse rate and temperature. Clinically significant changes in vital signs were to be reported as adverse events.
Time Frame: 16 weeks
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 14
participants | 0

ADVERSE EVENTS:
Time Frame: The time frame for adverse event (AE) reporting was up to 16 weeks and comprised the time from giving written informed consent (during screening) to 28 days after the last administration of study treatment.
Arm/Group | FXIII
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 8/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FXIII (N=14)
Acute bronchitis (Infections and infestations) | 2 (2)
Flu (Infections and infestations) | 1 (1)
Infected sebaceous cyst (Infections and infestations) | 1 (1)
Tinea corporis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle injury (Injury, poisoning and procedural complications) | 1 (1)
Bruising of arm (Injury, poisoning and procedural complications) | 1 (1)
Contusion of knee (Injury, poisoning and procedural complications) | 1 (1)
Contusion of toe (Injury, poisoning and procedural complications) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1)
Prothrombin increased (Investigations) | 1 (1)
Thrombin-antithrombin III complex increased (Investigations) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Borderline diabetes (Metabolism and nutrition disorders) | 1 (1)
Penile adhesion (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to public release. The sponsor may request any changes necessary to prevent forfeiture of patent rights to data not in the public domain. For a multi-center study, the investigator must wait (i) at least 1 year after the study is completed at all sites or (ii) until notified by the sponsor that no multi-center publication is planned, before seeking publication review.